CLINICAL TRIAL: NCT04983030
Title: A Safety, Immunogenicity and Efficacy Phase 1/2a Study of a Heterologous Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Regimen Plus Broadly Neutralizing Antibodies PGT121, PGDM1400, and VRC07-523LS in HIV-1-Infected Adults on Suppressive ART
Brief Title: Safety, Immunogenicity, Efficacy of Ad26.Mos4.HIV, MVA-BN-HIV and PGT121, PGDM1400, and VRC07-523LS in HIV-1-Infected Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boris Juelg, MD PhD (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Harvard School of Public Health (HSPH) (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Boris Juelg, MD PhD, Physician, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPCAVD014/HTX1004; 5U01AI145801 (NIH); 38743 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2021-07-05; First posted 2021-07-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome; Immunologic Deficiency Syndrome, Acquired; Sexually Transmitted Diseases, Viral; Retroviridae Infections
Keywords: Monoclonal antibodies; Therapeutic vaccination; Analytical treatment interruption; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases, Viral; Retroviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus PGT121, PGDM1400, and VRC07-523LS bNAbs (Experimental): Participants will receive Ad26.Mos4.HIV vaccine at week 0 and MVA-BN-HIV vaccine at week 12. The bNAbs PGT121, PGDM1400, and VRC07-523LS will be administered at week 24, and the bNAbs PGT121 and PGDM1400 will be administered at week 28.
  Interventions: Biological: Ad26.Mos4.HIV; Biological: MVA-BN-HIV; Biological: PGT121; Biological: PGDM1400; Biological: VRC07-523LS
- Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus Placebo (Active Comparator): Participants will receive Ad26.Mos4.HIV vaccine at week 0 and MVA-BN-HIV vaccine at week 12. Placebo will be administered at week 24, and at week 28.
  Interventions: Biological: Ad26.Mos4.HIV; Biological: MVA-BN-HIV
- Placebo Plus PGT121, PGDM1400, and VRC07-523LS bNAbs (Active Comparator): Participants will receive Placebo at week 0 and 12. The bNAbs PGT121, PGDM1400, and VRC07-523LS will be administered at week 24, and the bNAbs PGT121 and PGDM1400 will be administered at week 28.
  Interventions: Biological: PGT121; Biological: PGDM1400; Biological: VRC07-523LS

INTERVENTIONS:
Biological: Ad26.Mos4.HIV — Ad26.Mos4.HIV is a tetravalent vaccine containing Mos1.Env, Mos2S.Env, Mos1.Gag-Pol, and Mos2.Gag-Pol HIV-1 proteins.
  Arms: Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus PGT121, PGDM1400, and VRC07-523LS bNAbs; Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus Placebo
Biological: MVA-BN-HIV — MVA-BN-HIV is a monovalent vaccine comprising a single Modified Vaccinia Ankara - Bavarian Nordic (MVA-BN®) vector encoding Mos1.Env, Mos2S.Env, Mos1.Gag-Pol, and Mos2.Gag-Pol HIV-1 proteins.
  Arms: Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus PGT121, PGDM1400, and VRC07-523LS bNAbs; Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus Placebo
Biological: PGT121 — PGT121 is a human mAb that targets the HIV-1 V3 glycan, centered on N332.
  Arms: Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus PGT121, PGDM1400, and VRC07-523LS bNAbs; Placebo Plus PGT121, PGDM1400, and VRC07-523LS bNAbs
Biological: PGDM1400 — PGDM1400 is a human mAb that targets the HIV-1 V2 glycan, centered on N160.
  Arms: Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus PGT121, PGDM1400, and VRC07-523LS bNAbs; Placebo Plus PGT121, PGDM1400, and VRC07-523LS bNAbs
Biological: VRC07-523LS — VRC-HIVMAB075-00-AB (VRC07-523LS) is a human monoclonal antibody (mAb) that targets the HIV-1 CD4 binding site.
  Arms: Ad26.Mos4.HIV, MVA-BN-HIV Vaccine Plus PGT121, PGDM1400, and VRC07-523LS bNAbs; Placebo Plus PGT121, PGDM1400, and VRC07-523LS bNAbs

SUMMARY:
A multicenter, randomized, parallel-group, placebo-controlled, double-blind, Phase 1/2a clinical study to investigate the safety, tolerability, immunogenicity and exploratory efficacy of a vaccine regimen consisting of an Ad26.Mos4.HIV prime and a boost with Modified Vaccinia Ankara (MVA)-BN-HIV in combination with broadly neutralizing antibodies (bNAb) PGT121, PGDM1400, and VRC07-523LS in human immunodeficiency virus type 1 (HIV-1)-infected study participants on suppressive anti-retroviral therapy (ART).

DETAILED DESCRIPTION:
The study will enroll 36 adults randomized in a 1:1:1 ratio to 3 groups (vaccines+ bNAbs, vaccine+placebo, placebo+bNAbs), respectively. The study population will include HIV-infected adults who are on suppressive ART for at least 48 weeks prior to screening. The study comprises of a screening period of 10 weeks (Stage 0), a 24-week vaccination and follow-up period (Stage 1), a 4-week bNAb administration period and a 20-week bNAb washout period (Stage 2), and a 24-week monitoring period (Stage 3). An analytical antiretroviral treatment interruption (ATI) to assess rates of sustained virologic suppression will be conducted during Stages 2-3. Participants will record solicited signs and symptoms in a diary on the evening after each study drug administration and then daily for the next 7 days. Further safety evaluations will include monitoring of AEs, physical examinations, vital sign measurements, clinical laboratory tests (including urinalysis, CD4 count and HIV RNA), and for women, also pregnancy testing. Blood samples will be taken at specific clinic visits to assess immune and virologic responses as well as the pharmacokinetics and pharmacodynamics of bNAbs.

ELIGIBILITY:
Inclusion Criteria:

1. Each potential study participant must pass the Test of Understanding (TOU), indicating that he or she understands the purpose of, and procedures required for the study, after reading the informed consent and after the investigator or designee has provided detailed information on the study and has answered the potential study participant's questions. Each study participant must subsequently sign the ICF, indicating that he or she is willing to participate in the study.
2. Each study participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
3. Study participants are ≥18 to ≤70 years old on the day of signing the ICF.
4. Each study participant must have documented HIV-1 infection.
5. Must be on suppressive ART for at least 48 weeks prior to screening. ART is defined as a combination therapy regimen including at least 2 compounds, e.g., integrase inhibitor and nucleoside reverse transcriptase inhibitors (such as DovatoTM) or more than 2 compounds, e.g., 2x nucleoside reverse transcriptase inhibitors plus integrase inhibitor.
6. Must have a plasma HIV RNA <50 cps/mL at screening and at least 1 documented evidence of plasma HIV RNA <50 cps/mL after the last ART change.
7. Must be willing to undergo ATI.
8. Must be medically stable as confirmed by medical history, physical examination, vital signs, and clinical laboratory tests performed at screening, and as per the investigator's discretion.
9. Ability and willingness to restart ART according to study guidelines.
10. Each study participant must meet the following laboratory criteria prior to randomization:

    * Hemoglobin: Women ≥10.5 g/dL; Men ≥11.0 g/dL
    * White cell count: 2,500 to 11,000 cells/mm3, inclusive
    * Absolute neutrophil count: >1,000 cells/mm3
    * Platelets: 125,000 to 450,000 per mm3, inclusive
    * Screening serum liver enzymes (e.g., alanine aminotransferase [ALT], aspartate aminotransferase [AST], total bilirubin): within the normal reference ranges at baseline
    * Creatinine: <1.2 x ULN
    * Estimated glomerular filtration rate ≥ 60 mL/min
    * CD4+: >450 cells/mm3 at screening and at least 1 documented result >300 cells/mm3 during 48 weeks before randomization (for nadir, see exclusion criterion 9)
    * Troponin: <1 x ULN
11. For participants who are able to become pregnant, negative serum or urine pregnancy test (with a sensitivity of 15-25 mIU/mL) within 24 hours prior to Stage 1 randomization
12. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction starting from the first vaccination at Week 0 visit and for a period of 24 weeks after last dose of bNAb.

Exclusion Criteria:

1. Anyone who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study.
2. Anyone with contraindication to intramuscular injections, placement of intravenous lines, and blood draws eg, bleeding disorders. NOTE: nonsteroidal anti- inflammatory drugs (NSAIDS) and acetylsalicylic acid containing preparations have to be stopped for 5 days before and after planned leukapheresis.
3. Anyone with acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature ≥38.0oC within 24 hours prior to the first dose of study vaccine; enrollment at a later date is permitted.
4. Any history of an HIV-associated malignancy (including Kaposi's sarcoma), and any type of lymphoma, or virus-associated cancers.
5. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the 36 months prior to Stage 1 randomization or for whom such therapies are expected in the next 12 months (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence).
6. Anyone with a history of an underlying clinically significant acute or uncontrolled chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the study participant.
7. History or current clinical atherosclerotic cardiovascular disease, as defined by 2013 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines, including a previous diagnosis of any of the following:

   * Acute myocardial infarction
   * Acute coronary syndromes
   * Stable or unstable angina
   * Coronary or other arterial revascularization
   * Stroke
   * TIA
   * Peripheral arterial disease presumed to be of atherosclerotic origin
8. Anyone with a history of HIV-related illness under CDC Category C (except for recurrent pneumonia) within 10 years prior to screening, based on available medical history and assessed by the investigator for clinical relevance.
9. Anyone with a history of repeated CD4+ <200 cells/mm3, based on available medical history and assessed by the investigator for clinical relevance. .
10. Current receipt of ART other than nucleoside reverse transcriptase inhibitor and integrase inhibitor.
11. Anyone who had major surgery (per the investigator's judgment), within 12 weeks before dosing, or has not have fully recovered from surgery, or has surgery planned during the time the study participant is expected to participate in the study or within 6 months after the last dose of study vaccine administration.
12. Anyone with a history of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up).
13. Anyone with an ECG with reading and showing clinically significant findings, or features that would interfere with the assessment of myocarditis/pericarditis.
14. Current advanced liver disease (non-alcoholic fatty liver disease, steatohepatitis, or alcoholic liver disease) with known or suspected cirrhosis or fibrosis score ≥F2.
15. Anyone with chronic active hepatitis B (measured by hepatitis B surface antigen test) or active hepatitis C (measured by hepatitis C virus [HCV] antibody test; if positive, HCV RNA polymerase chain reaction test will be used to confirm active versus past HCV infection) or syphilis infection that has not been effectively treated. Positive syphilis serology due to past effectively treated infection is not exclusionary.
16. Anyone with active, untreated gonorrhea or chlamydia infection will be referred to a clinician for appropriate treatment. If chlamydia and/or gonorrhea treatment is successfully completed, the participant is eligible for a repeat gonorrhea or chlamydia screening test and potential study entry.
17. Anyone with thyroidectomy or active thyroid disease requiring medication during the last 12 months (Not excluded: a stable thyroid supplementation).
18. Anyone with history of HIV-associated neurocognitive disease or progressive multifocal leukoencephalopathy.
19. Anyone who has had major psychiatric illness and/or drug or alcohol abuse which in the investigator's opinion would compromise the study participant's safety and/or compliance with the study procedures.
20. Anyone with a history of thrombosis with thrombocytopenia syndrome (TTS), or Heparin-induced thrombocytopenia and thrombosis syndrome (HITTS)
21. Anyone who received treatment with immunoglobulins in the 2 months or blood products in the 4 months before the planned administration of the first dose of study vaccine or has any plans to receive such treatment during the study. Prior recipients of anti-HIV bNAbs, independently of the timing, are excluded.
22. Anyone who received or plans to receive:

    1. licensed live attenuated vaccines - within 28 days before or after planned administration of any of the study products.
    2. other licensed (not live) vaccines - within 14 days before or after planned administration of any of the study products.
    3. SARS-CoV-2 vaccines under Emergency Use Authorization (EUA) by the FDA - within 28 days before or after planned administration of any of the study products.
23. Anyone who received an investigational drug (not under EUA by the FDA) or used an invasive investigational medical device within 30 days or received an investigational vaccine within 6 months before the planned administration of the first dose of study vaccine. Receipt of prophylactic or therapeutic HIV vaccine candidate at any time is always exclusionary.
24. Anyone who is currently enrolled or plans to participate in another investigational study during the course of this study.
25. Anyone who has known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines) and specifically to neomycin or streptomycin or egg products.
26. Anyone with a history of chronic urticaria (recurrent hives) or a history of chronic or recurrent eczema and/or atopic dermatitis.
27. Anyone with abnormal function of the immune system resulting from:

    1. Clinical conditions (e.g., autoimmune disease or immunodeficiency that are not HIV related).
    2. Chronic or recurrent use of systemic corticosteroids.
    3. Administration of antineoplastic and immunomodulating agents or radiotherapy.
28. Anyone with history of acute polyneuropathy(e.g.,Guillain-Barré syndrome).
29. Anyone who cannot communicate reliably with the investigator.
30. Known resistance to 1 or more drugs in 2 or more ARV drug classes.
31. Weight >115kg.
32. Anyone who, in the opinion of the investigator, is unlikely to adhere to the requirements of the study, or is unlikely to complete the full course of vaccination and observation.
33. Any employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator, or an employee of the sponsor (or its partners).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Solicited Local Adverse Events (AEs) as a Measure of Safety and Tolerability | 7 days post-investigational product administration
  Solicited local AEs: erythema, swelling/induration, and pain/tenderness will be assessed.
Percentage of Participants With Solicited Systemic AEs as a Measure of Safety and Tolerability | 7 days post-investigational product administration
  Solicited systemic AEs: fever (temperature measurement), fatigue, headache, nausea, myalgia, and chills will be assessed.
Percentage of Participants With Unsolicited AEs as a Measure of Safety and Tolerability | Approximately up to 72 weeks
  An Unsolicited AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Percentage of Participants With Adverse Events of Special Interest (AESIs) | From first vaccination until 6 months after last vaccination.
  AESIs and potential AESIs are judged to be of special interest because of clinical importance, known or suspected class effects and include thrombotic events and symptomatic thrombocytopenia.
Frequency of Epitope Recognition by Enzyme-Linked Immunospot (ELISPOT) | Up to post-vaccination follow-up period until Week 72
  Assays of peptide pool sets covering the Gag, Env or Pol will be evaluated by standard enzyme linked immunospot assay (ELISPOT).
Total IgG and Subclass Specific Antibody Titer | Up to post-vaccination follow-up period until Week 72 ]
  Total immunoglobulin G (IgG) and subclass (IgG1-4) specific antibody titers (binding antibody) to envelope (Env) proteins representing Clades A, B, and C, as well as Mosaic antigens.
Antiviral activity - Percentage of participants who maintain plasma HIV RNA <1000 copies/mL | Time between week 24 and week 72 week
  Proportion of participants who remain off ART and maintaining plasma HIV RNA <1000 copies/mL for at least two thirds of the time between 24 and 72 weeks of analytical treatment interruption (ATI).

SECONDARY OUTCOMES:
Measurement of the HIV-1 reservoir (dQVOA) | At baseline, Week 24 and Week 32
  Measurement of the HIV-1 reservoir by differential quantitative viral outgrowth assay
Measurement of intact proviral DNA | At baseline, Week 24 and Week 32
  Measurement of intact proviral DNA, ie by intact proviral DNA assay (IPDA)
Compare the time to viral rebound (defined as confirmed plasma HIV RNA levels ≥1,000 copies/mL) following Ad26.Mos4.HIV, MVA-BN-HIV and placebo with the results of the rates of viral rebound as observed in historical controls. | Week 48
  The proportion of participants in Group 2 who remain off ART maintaining plasma HIV RNA <1000 cps/mL at Week 48 compared to historical controls
To evaluate PGT121, VRC07-523LS and PGDM1400 serum levels at which viral rebound is detected during the analytical treatment interruption. | From start of ATI until the date of HIV RNA >1000 copies/ml assessed up to week 72
  Serum levels of PGT121, VRC07-523LS and PGDM1400 at time of viral rebound.
HIV genotyping of circulating virus | From start of ATI until the date of HIV RNA >1000 copies/ml assessed up to week 72
  Genotypic analysis: Development of sequence variations in epitopes known to result in reduced PGDM1400 mAb and/or PGT121 mAb and/or VRC07-523LS mAb neutralization susceptibility
HIV phenotyping of circulating virus | From start of ATI until the date of HIV RNA >1000 copies/ml assessed up to week 72
  Phenotypic analysis: Changes in viral susceptibility to PGDM1400 mAb and/or PGT121 mAb and/or VRC07-523LS mAb neutralization

CONTACTS AND LOCATIONS:
Overall Officials: Boris D Juelg, MD PHD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (6):
- United States (6):
  - UCLA CARE (Center for AIDs Research and Education), Los Angeles, California
  - Orlando Immunology Center, Orlando, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University Clinical Trials Unit, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Washington Positive Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all IPD that underlie the results reported in a respective publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.